CLINICAL TRIAL: NCT04964284
Title: A Randomized, Open-label, Multi-center, Controlled Phase Ⅲ Study to Evaluate the Safety and Efficacy of Recombinant Human Thryoid Stimulating Hormone（rhTSH） for Adjuvant Radioiodine Ablation Therapy in Postoperative Patients With Differentiated Thyroid Cancer
Brief Title: Efficacy and Safety Study of rhTSH for Adjuvant Radioiodine Ablation Therapy in Patients With Differentiated Thyroid Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGTSH003
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — Thyrotropin Alfa; Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTSH group (Experimental): Patients received thyroid hormone suppression therapy (Euthyrox) . rhTSH (0.9 mg) was administered intramuscularly (IM) once daily (qd) for 2 days. Twenty-four hours following the second dose of rhTSH, an ablative activity of 131I (30 mCi±1.5 mCi) was administered.
  Interventions: Biological: rhTSH; Radiation: Radioiodine (131I)
- Thyroid hormone withdrawal group (Experimental): After randomization, patients with thyroid hormone withdrawal therapy(i.e. Stop taking thyroid hormone for 14 days, and then monitor the level of thyroid-stimulating hormone every week). When TSH>30mU/L, an ablative activity of 131I (30 mCi±1.5 mCi) was administered.
  Interventions: Radiation: Radioiodine (131I)

INTERVENTIONS:
Biological: rhTSH — rhTSH (0.9 mg) was administered intramuscularly (IM) once daily (qd) for 2 days. Twenty-four hours following the second dose of rhTSH
  Other Names: Recombinant human thyroid-stimulating hormone
  Arms: rhTSH group
Radiation: Radioiodine (131I) — Patients were given an ablative dose of 131I (30 mCi±1.5 mCi).

SUMMARY:
This study was conducted in patients with differentiated thyroid cancer who had undergone total/near-total thyroidectomy. After surgery patients were randomized to one of two methods of performing thyroid remnant ablation. One group of patients who took thyroid hormone medicine and were euthyroid [i.e. their thyroid stimulating hormone (TSH) levels are normal], and received injections of rhTSH (0.9 mg daily on two consecutive days) followed by oral radioiodine. The second group of patients did not take thyroid hormone medicine so that they were hypothyroid (i.e. their TSH levels were high), and were given oral radioiodine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily sign the informed consent form (ICF).
* Age ≥ 18 years old, either male or female.
* Patients with diagnosed differentiated papillary or follicular thyroid carcinoma, including papillary-follicular variant, characterized as pT 1-3, N 0-1or Nx, and M0.
* Eastern Cooperative Oncology Group (ECOG) score of 0-2;
* Expected life expectancy is greater than 12 weeks;
* Patients with a total or near-total thyroidectomy within 12 months prior to randomized.
* Low iodine diet for two weeks prior to randomized.

Exclusion Criteria:

* patients with recent history of 131I whole body scan within 2 weeks prior to randomized.
* Pregnant or breast feeding women.
* patients with other malignancies (exception for in situ cervix uterine cancer, baso cellular skin cancer or breast cancer in remission)
* Subjects who are unsuitable to the trial in combination with other serious diseases, as identified by the investigator.
* Subjects who have participated in another clinical trial of a new drug or medical instrument within 1 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The rate of successful postoperative thyroid ablation | 8 months later by a rhTSH stimulated radioiodine scan
  Patients were considered successfully ablated if there was no visible thyroid bed uptake on the scan

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Lin, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China